# **Evaluating the Social Workers Addressing Firearm Risk (SAFR) Intervention: A Pilot Study Informed Consent Information**

## January 31, 2023

This pilot study is being conducted by Patricia Logan-Greene, PhD; Mickey Sperlich, PhD; and Gregory Wilding, PhD, researchers from the University at Buffalo. This research is funded by the Clinical and Translational Science Institute at the University at Buffalo.

This study entails a randomized controlled trial to evaluate the preliminary efficacy of Social Workers Addressing Firearm Risk (SAFR) Intervention, an online course to train practicing social workers on understanding, recognizing, and responding to risks of firearm violence injury among their clients. The online course is self-paced and takes about six hours to complete within 30 days. We expect about 100 social workers to be part of this study.

#### Why am I being invited to participate in this study?

You are being invited to take part in this research study because you are a practicing social worker. Participation in research is completely voluntary. You can ask all the questions you want before you decide. You may choose not to enroll in this study. Your alternative to participating in this research study is to not participate. You can agree to take part and later change your mind, and your decision will not be held against you. Although unlikely, the person in charge of the research study or the sponsor can remove you from the research study without your approval.

#### What will happen if I agree to participate in this study?

Participation in this study includes completing an initial questionnaire about your firearm knowledge, attitudes, beliefs, and behaviors with your clients, which will take about 20-30 minutes to complete. Participants will then be sorted randomly into two groups: an intervention and control group. If you are placed in the intervention group, you will receive access to the online course. You will have 30 days to complete the self-paced 6-hour course. If eligible based on clinical certification, you will receive 6 continuing education units upon completing the course. One month after completion, you will receive a post-test (similar to the first questionnaire, and which will also take about 20 minutes to complete) and two months after that, you will receive a follow-up test (again, 20 minutes).

If you are placed in the control group, you will receive the pre, post, and follow-up tests on the same timeline as above, but not the SAFR course materials. You will be given free access to the SAFR course upon completion of the study.

All communications and questionnaires will occur by email. If you take part in this research, you will be responsible for answering all questions honestly and completing questionnaires in a timely manner.

# Are there risks to participating in this study?

The information in the SAFR course and the questions in the questionnaires are related to firearms and firearm violence. The risk of harm is minimal, but the content could make you feel uncomfortable, upset, or offended if you have experienced an adverse event related to firearms. If you experience an adverse reaction, help is available by calling "988," which is a crisis hotline that provides 24/7, free and confidential support for people in distress across the United States.

There is a small chance that someone who is not authorized could see your private study information. We are taking steps so that does not happen. Efforts will be made to limit the use and disclosure of your personal information, including your email addresses and research study records, to people who have a need to review this information. All study documents will be stored on secure University at Buffalo servers that are only accessible to research team members on password-protected computers. We cannot promise complete secrecy. Organizations that may inspect and copy your information

include the IRB and other representatives. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the study results. You can search this website at any time. Questionnaires will be submitted confidentially and be electronically stored with no identifiable information besides your email address.

Your data will be retained after the study for future research. Data will be stored in a data cloud hosted by University at Buffalo. Usernames and passwords are required to access the cloud and data information files will only be shared with members of the research team. Your data will be retained if you withdraw from the study unless you request that it be removed.

### What are the benefits from participating in this study?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include knowledge and skills that may help you reduce risk of firearm violence among your clients and create safer communities. Your participation could contribute to an increase in skills and knowledge social workers can utilize to address firearm violence.

For those who are eligible, completing the SAFR training will entitle you to six hours of continuing education credits through the University at Buffalo School of Social Work Continuing Education department. Those in the control group will receive access to the course and this credit at the end of the study.

If you have questions, concerns, or complaints, or think the research has hurt you, you can reach a study representative by emailing <a href="mailto:safrstudy@buffalo.edu">safrstudy@buffalo.edu</a>. You may also contact the research participant advocate at 716-888-4845 or <a href="mailto:researchadvocate@buffalo.edu">researchadvocate@buffalo.edu</a>.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). An IRB is a committee that provides ethical and regulatory oversight of research that involves human subjects. You may talk to them at (716) 888-4888 or email <a href="mailto:ub-irb@buffalo.edu">ub-irb@buffalo.edu</a> if:

- You have questions about your rights as a participant in this research
- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You want to get information or provide input about this research.

What happens if I say yes, I want to be in this research?

- You will be directed to a link to complete the initial questionnaire.
- You will have 7 days to complete the online questionnaire including your demographic questions.
- After all questions are answered, submit the questionnaire, and the information will be received by the research team.
- If you are assigned to the intervention group, you will obtain access to the SAFR course and have 30 days to complete it, submit a course evaluation, and receive the continuing education units.
- If you are in the control group, you will receive an email advising you of this. You will gain access to the course after the study is completed.
- One month after completing the first questionnaire, you will receive an additional link and complete the second questionnaire.
- Three months after completing the first questionnaire, you will receive an additional link to complete the final questionnaire.

If you agree to take part in this research study, we will pay you a \$30 gift card for completing the initial questionnaire, \$40 gift card for completing the second questionnaire one month later, and \$50

for completing the final questionnaire. You will also receive 6 hours of continuing education units upon successful completion of the SAFR course.

The Study Card Program Group, under The University at Buffalo Office of Financial Management, in conjunction with U.S. Bank, will manage study compensation by providing a One-Time Digital Reward Card. When you complete a study questionnaire, the amount outlined in the Informed Consent Form will be automatically approved and applied to your digital reward. The Study staff will provide you with additional information about how the digital reward card works. In order for U.S. Bank to be able to reimburse you using the One-Time Digital Reward Card, your email address will be collected and provided to U.S. Bank. The Study Card Program Group, under The University at Buffalo Office of Financial Management, will also have access to this information and UB affiliated Researchers and staff, within the same university department as the Investigator of this study, may also have access to this information. By agreeing to use the U.S. Bank Card service, you are authorizing the release of this information to U.S. Bank and authorizing access to this information to the Study Card Program Group, under The University at Buffalo Office of Financial Management and other UB affiliated Researchers and staff.

Please note that U.S. Bank may use your personal contact information to market the bank's other products and services to you. You may limit U.S. Bank's direct marketing to you by visiting U.S. Bank online at <a href="http://www.usbank.com/privacy">http://www.usbank.com/privacy</a>.

| By clicking on the continue button below, you are agreeing to participate in this study: | |
|---|---|
| I agree to participate in this study. | |
| I do not wish to participate in this study. | |
| Please provide your email here if you would like a copy of this consent form sent to you. (Optional | ) |